CLINICAL TRIAL: NCT04251013
Title: Multicenter RCT Comparing Two Brushes of Different Diameters for Biliary Stenosis: RX Cytology Brush, BOSTON vs. Infinity® Brush, US Endoscopy. BIB Study (BIliary Brushing)
Brief Title: Multicenter RCT for BIliary Brushing: RX Cytology, BOSTON vs. Infinity®, US Endoscopy
Acronym: BIB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, Principal Investigator, Société Française d'Endoscopie Digestive
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: BIB study
Record Dates: First submitted 2020-01-25; First posted 2020-01-31 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Biliary Stricture; Jaundice, Obstructive
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Intervention Model Description: National prospective multicenter RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: RX Cytology brush, Boston Scientific FIRST (Active Comparator): A first biliary brushing will be carried out during ERCP using a standard brush RX Cytology Brush, Boston Scientific, then a second brushing will be carried out using a brush INFINITY®, US Endoscopy
  Interventions: Device: Biliary brushing with the RX Cytology brush, Boston Scientific; Device: Biliary brushing with the Infinity® brush, US Endoscopy
- Group B: Infinity®, US Endoscopy FIRST (Active Comparator): A first biliary brushing will be carried out during ERCP using an INFINITY® brush, US Endoscopy then a second brushing will be carried out using standard RX Cytology Brush, Boston Scientific
  Interventions: Device: Biliary brushing with the RX Cytology brush, Boston Scientific; Device: Biliary brushing with the Infinity® brush, US Endoscopy

INTERVENTIONS:
Device: Biliary brushing with the RX Cytology brush, Boston Scientific — Biliary brushing during ERCP:
  * Performing a dozen back and forth movements in the stenosis
  * Bile aspiration if possible, by the catheter of the brush for cytological analysis
  * The contents of the brush will be spread over 3 blades (numbered) then sectioned and placed in cytolit with the contents of the tubing of the brush flushed with a few cc of cytolit. Each brush in a numbered pot. Blades 1,2 and 3 +/- bile 1 joined to pot n ° 1; blades 4,5 and 6 +/- bile 2 joined to pot 2
    * In the event of technical failure (impossibility of accessing the stenosis with the first or second brush, impossibility of removing the brush), the patient will be considered to have failed for this brush (absence of pathological material brought back)
Device: Biliary brushing with the Infinity® brush, US Endoscopy — Biliary brushing during ERCP:
  * Performing a dozen back and forth movements in the stenosis
  * Bile aspiration if possible, by the catheter of the brush for cytological analysis
  * The contents of the brush will be spread over 3 blades (numbered) then sectioned and placed in cytolit with the contents of the tubing of the brush flushed with a few cc of cytolit. Each brush in a numbered pot. Blades 1,2 and 3 +/- bile 1 joined to pot n ° 1; blades 4,5 and 6 +/- bile 2 joined to pot 2
    * In the event of technical failure (impossibility of accessing the stenosis with the first or second brush, impossibility of removing the brush), the patient will be considered to have failed for this brush (absence of pathological material brought back)

SUMMARY:
The aim of this prospective national multicenter randomized study is to compare, during an ERCP for VBP stenosis, the sensitivity of two biliary brushes: the INFINITY® vs the RX Cytology Brush® The main objective is the comparison of the rates of positive diagnosis of biliary brushing in cases of adenocarcinoma stenosis The total number of subjects required: 50 (25 patients per group) Duration of the inclusion period: 2 years Duration of participation for each subject: from 7 days to 12 months (in case of negative initial withdrawal) Total duration of the study: 3 years

DETAILED DESCRIPTION:
The aim of this study is to compare, during an ERCP for VBP stenosis, the sensitivity of two biliary brushes: the INFINITY® vs the RX Cytology Brush®

OBJECTIVES

* Main objective: Comparison of the rates of positive diagnosis of biliary brushing in cases of adenocarcinoma stenosis
* Secondary objective (s):

  * Comparison of the quantification of the cellular material obtained (acellular, weak, or abundant), and the presence of cellular cupboards unhooked by the brush
  * Comparison of the 2 brushes false negative rates, and negative predictive value for the diagnosis of adenocarcinoma
  * Evaluation of the variation in the profitability of brushing and other sampling techniques (intra-biliary biopsies, puncture, aspiration of bile) according to the presence of a tumor mass syndrome of more than 1 cm.
  * Evaluation of the variation in the profitability of brushing and other sampling techniques (intra-biliary biopsies, puncture, aspiration of bile) according to the site of the stenosis (distal vs proximal BPV: common bile duct or intrahepatic duct), with the cost effectiveness
  * Technical failure rate of brushing and other samples (intra-biliary biopsies, bile aspiration)

This study concerns adult subjects with stenosis of the main bile duct (common bile duct or common hepatic duct).

ENDOSCOPIC PROCEDURE

* Deep catheterization of the biliary duct (whatever the access technique: by the papilla or by precut) and cross stenosis by the guide wire, then biliary dilation (6 to 8mm)
* Randomization if the inclusion criteria are met
* Biliary brushing successively with the 2 brushes in the order designated by randomization:

  * Performing a dozen back and forth movements in the stenosis
  * Aspiration, if possible of bile by the catheter of the brush for cytological analysis
  * The contents of the brush will be spread over 3 blades (numbered) then sectioned and placed in cytolit with the contents of the tubing of the brush flushed with a few cc of cytolit. Each brush in a numbered pot. Blades 1,2 and 3 +/- bile 1 joined to pot n ° 1; blades 4,5 and 6 +/- bile 2 joined to pot 2
* In the event of technical failure (impossibility of accessing the stenosis with the first or second brush, impossibility of removing the brush), the patient will be considered to have failed for this brush (absence of pathological material brought back)

All possible sampling methods will also be taken to obtain the anatomopathological diagnosis: intra-biliary biopsies with adult or pediatric forceps, wire-guided or not, biopsy samples guided by choledochoscopy, puncture under endo-ultrasonography, bile aspiration after release of the biliary stent, according to the physician's habits.

EFFECTIVE The total number of subjects required: 50 (25 patients per group) Duration of the inclusion period: 2 years Duration of participation for each subject: from 7 days to 12 months (in case of negative initial withdrawal) Total duration of the study: 3 years

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to one of the ERCP investigation centers with brushing and drainage for VBP stenosis (proximal or distal) during the study period
* Patient whose age is greater than or equal to 18 years and less than 90 years
* Patient ASA 1, ASA 2, ASA 3
* Lack of participation in another clinical study
* Signed informed consent

Exclusion Criteria:

* Patients admitted for ERCP for jaundice by lithiasic obstruction
* Patient under 18 or over 90
* Patient ASA 4, ASA 5
* Pregnant woman
* Patient (s) with coagulation abnormalities preventing puncture: TP <50%, Platelets <50,000 / mm3, effective anti-coagulation in progress, clopidogrel in progress
* Surgical setup (Billroth II, Roux en Y) preventing endoscopic access to the papilla
* Patient unable to give personal consent
* Lack of signed informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Sensibility for adenocarcinoma | 8 days to 1 year (if negative)
  Rate of positive diagnosis of biliary brushing in case of cholangiocarcinoma stenosis

SECONDARY OUTCOMES:
Sample abundance | 8 days
  Quantification of the cellular material obtained (acellular, weak, or abundant), presence of cellular cupboards unhooked by the brush or average number of cells per field
False negative | 1 year
  Negative brushing for a final diagnosis of cholangiocarcinoma
Predictive Negative Value | 1 year
  probability that patients with a negative brushing truly don't have cholangiocarcinoma
Feasibility of the 2 brushes: Analog visual scale | 1 day
  Analog visual scale: Feasibility scale (0 to 10, 0 for Extremely difficult to perform and 10 for very easy to perform)
Feasibility of the intra-biliary biopsies: Analog visual scale | 1 day
  Analog visual scale: Feasibility scale (0 to 10, 0 for Extremely difficult to perform and 10 for very easy to perform)
Feasibility of bile aspiration: Analog visual scale | 1 day
  Analog visual scale: Feasibility scale (0 to 10, 0 for Extremely difficult to perform and 10 for very easy to perform)
Feasibility of stenosis puncture under ultrasonography: Analog visual scale | 1 day
  Analog visual scale: Feasibility scale (0 to 10, 0 for Extremely difficult to perform and 10 for very easy to perform)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Paris Bercy, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karsenti D, Privat J, Charissoux A, Perrot B, Leblanc S, Chaput U, Boytchev I, Levy J, Schaefer M, Bourgaux JF, Valats JC, Coron E, Moreno-Garcia M, Vanbiervliet G, Rahmi G, Robles EP, Wallenhorst T. Multicenter randomized trial comparing diagnostic sensitivity and cellular abundance with aggressive versus standard biliary brushing for bile duct stenosis without mass syndrome. Endoscopy. 2023 Sep;55(9):796-803. doi: 10.1055/a-2041-7687. Epub 2023 Feb 27. PMID 36849106